CLINICAL TRIAL: NCT06805071
Title: Decisional Regret in Open Partial Horizontal Laryngectomy
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: DROPHL-2023
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-05

CONDITIONS: Laryngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Prospective multicentric study to evaluate decisional regret and psychometric and functional outcomes in patient previously treated with Open Horizontal partial Laryngectomy

ELIGIBILITY:
Inclusion Criteria:

* SCC larynx treated with OPEN PARTIAL HORIZONTAL LARYNGECTOMY

Exclusion Criteria:

* Previous surgical treatment of the larynx
* Previous CT-RT of the head and neck district

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with laryngeal squamous cell carcinoma of any stage amenable of organ preservation surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-01-25 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Decisional Regret Scale | From the surgery to the enrollment time (6 months post-treatment)
  Evaluation of subjective regret about the therapeutic choice

SECONDARY OUTCOMES:
DASS-21 Questionnaire | From the surgery to the enrollment time (6 months post-treatment)
  21 items-questionnaire about depression, anxiety and stress during the post-treatment period
Chicago Priority Scale | From the surgery to the enrollment time (6 months post-treatment)
  12 items-ranking of Oncological therapeutic objectives of the Head and Neck patient
VHI-10 | From 6 Months after surgery until the end of the study
  Self evaluation of the dysphonia after surgery
MD Anderson Dysphagia Inventory | From 6 Months after surgery until the end of the study
  Self evaluation of dysphagia post surgical treatment + adjuvant therapy if administered

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Fermi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, BO, Italy